CLINICAL TRIAL: NCT01088139
Title: A Randomized Controlled Study of Nutritional Intervention for Geriatric Hip Fracture Patients and Its Effect on Rehabilitation Outcomes
Brief Title: Nutritional Intervention for Geriatric Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Responsible Party: Dr MYINT Ma Wai Wai, Associate Consultant, Department of Rehabilitation, Kowloon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KC/KE-08-0118/ER3
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: Hip Fractures
Keywords: Nutritional support; Rehabilitation outcomes
MeSH Terms: conditions — Hip Fractures | interventions — Glucerna

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Nutritional Supplementation (Experimental)
  Interventions: Dietary Supplement: Protein supplementation

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Ready made protein supplement drinks with approximate protein content of 18-24g per 500ml per day. Caloric content is 490 to 530Kcal depending on the brand of drink.
  Other Names: Ensure (Abbott); Resource Breeze (Nestle Nutrition); Compleat (Nestle Nutrition); Glucerna (Abbott)
  Arms: Nutritional Supplementation

SUMMARY:
This is a randomized controlled, observer blinded trial to study the beneficial effect of nutritional supplementation in elderly Hong Kong patients after hip fracture surgery during rehabilitation and at 4 weeks follow up. The control group will receive Calcium and Vitamin D supplementation whereas the intervention group will receive a moderately high dose protein nutritional supplementation in addition to Vitamin D and Calcium. Both groups undergo the same rehabilitation program and dietary counseling before discharge. They are followed up 4 weeks after discharge or completion of supplementation. The outcome parameters are nutritional parameters and rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Recent low impact osteoporotic fracture of the proximal femur surgically repaired within 4 weeks before recruitment

Exclusion Criteria:

* Patients who require tube feeding
* Patients in unstable medical condition
* Body mass index (BMI) ≧ 25
* Malignancy
* Conditions with contraindication for high protein diet
* Mentally incapacitated and inability to communicate or understand the consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Nutritional parameters | Change from Baseline in nutritional parameters at discharge from hospital and at 4 weeks after discharge
  Biochemical and anthropometric measurements

SECONDARY OUTCOMES:
Rehabilitation Outcomes | Change from Baseline in rehabilitation outcomes at discharge from hospital and at 4 weeks after discharge
  functional, strength and mobility measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ma Wai Wai MYINT, MBBS, Principal Investigator — Kowloon Hospital, Hong Kong
Locations (1):
- Department of Rehabilitation, Kowloon Hospital, Kowloon, Hong Kong